CLINICAL TRIAL: NCT07076758
Title: Correlation Between Serum Copper and Cardiac Enzymes in Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Remon Saleh Adly, Lecturer of Cardiovascular, Faculty of Medicine, Sohag University, Sohag, Egypt., Sohag University
Other Study IDs: Soh-Med-25-5-7PD
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Serum Copper; Cardiac Enzymes; Acute Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Patients with acute myocardial infarction.
  Interventions: Other: Transthoracic echocardiography
- Group II: Healthy control individuals as a control group.
  Interventions: Other: Transthoracic echocardiography

INTERVENTIONS:
Other: Transthoracic echocardiography — Transthoracic echocardiography will be done for all patients during their cardiac care unit stay including two-dimensional and color Doppler echocardiography studies. It will be performed in the left lateral position using the parasternal and apical transducer positions. All studies will be technically adequate for scoring endocardial regional wall motion. The following views will be obtained: long-axis parasternal, short-axis parasternal, apical four chamber, apical two-chamber and apical five-chamber views. All the measurements taken will be according to the criteria of the American Society of Echocardiography

SUMMARY:
This study aims to investigate the correlation between serum copper levels and cardiac enzymes in patients with acute myocardial infarction (AMI).

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is one of the most serious types of coronary artery disease (CAD). In CAD, coronary blood flow is drastically reduced or interrupted, causing severe myocardial ischemia or necrosis.

Cardiac troponin I (TNI), creatine kinase (CK), and creatine kinase MB (CK-MB) are the most commonly used biomarkers for AMI clinical diagnosis. Among them, cardiac troponin is a highly specific biomarker for the diagnosis of AMI. However, the sensitivity is not good in the first few AMI hours, and false-positive values may occur in severe heart failure, arrhythmia, and myocarditis.

Copper is vital in multiple enzymes necessary for antioxidant protection, such as Superoxide dismutases (SOD) and ceruloplasmin. SOD is an enzyme that changes superoxide radicals into hydrogen peroxide, whereas ceruloplasmin is an antioxidant protein that aids in eliminating free radicals.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Both sexes.
* Patients with acute myocardial infarction (AMI). AMI are defined as patients complaining of typical continuous chest pain for more than 30 min: ST-segment elevation of more than 0.1 mV in two or more successive leads or ST-segment depression of more than 0.1 mV in two or more successive leads monitored by a standard 12-lead ECG and rise of either creatine kinase (CK) or MB fraction of creatine kinase (CKMB) to greater than twice the normal level or elevation of troponin I [cardiac troponin T (cTnT)] more than or equal to 0.1 ng/ml

Exclusion Criteria:

* Patients with insufficient clinical information.
* Passed time MI (if patients presented with symptoms that lasted >24 h).
* Cardiogenic shock.
* Chronic kidney disease.
* Chronic liver cell failure.
* Significant valvular heart disease.
* Hematological disease.
* Malignancy.
* Severe liver or renal disease.
* Systemic inflammatory disease.
* Active infection.
* Autoimmune disease.
* Patients on steroids whatever the cause is.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This case-control study will be conducted at Sohag University Hospitals after approval from the institutional ethical committee.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Serum copper level | Immediately after echocardiography (Up to 1 hour)
  Serum copper level will be recorded.

SECONDARY OUTCOMES:
Correlation between copper zinc and cardiac enzyme | Immediately after echocardiography (Up to 1 hour)
  Correlation between copper zinc and cardiac enzyme will be done.
Creatine kinase | Immediately after echocardiography (Up to 1 hour)
  Creatine kinase level will be recorded.
MB fraction of creatine kinase | Immediately after echocardiography (Up to 1 hour)
  MB fraction of creatine kinase will be recorded.
Cardiac troponin T | Immediately after echocardiography (Up to 1 hour)
  Cardiac troponin T will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.